CLINICAL TRIAL: NCT00492167
Title: Phase I Study of Oral Yeast β-Glucan and Intravenous Anti-GD2 Monoclonal Antibody 3F8 Among Patients With Metastatic Neuroblastoma
Brief Title: Beta-Glucan and Monoclonal Antibody 3F8 in Treating Patients With Metastatic Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-073; MSKCC-05073
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — beta-Glucans; humanized 3F8 anti-GD2 monoclonal antibody; Immunohistochemistry

ARMS (1):
- Beta-Glucan and Monoclonal Antibody 3F8 (Experimental): This is a dose-escalation study of beta-glucan. Patients receive oral beta-glucan once daily on days -4 to 12 and monoclonal antibody 3F8 IV over 30-90 minutes on days 1-5 and 8-12. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity and with a human antimouse antibody (HAMA) titer < 1,000 U/mL.
  Cohorts of 3-6 patients receive escalating doses of beta-glucan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Patients undergo urine, bone marrow, and blood sample collection periodically for biological studies. Samples are analyzed for antibody-dependent cellular cytotoxicity, complement-mediated cytotoxicity, and serum HAMA response via immunohistochemistry.
  After completion of study treatment, patients are followed periodica
  Interventions: Biological: beta-glucan; Biological: monoclonal antibody 3F8; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: beta-glucan
Biological: monoclonal antibody 3F8
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Beta-glucan may stimulate the immune system and stop tumor cells from growing. Monoclonal antibodies, such as 3F8, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving beta-glucan together with monoclonal antibody 3F8 may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of beta-glucan when given together with monoclonal antibody 3F8 in treating patients with metastatic neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical toxicity of beta-glucan in combination with monoclonal antibody 3F8 in patients with metastatic neuroblastoma.
* Evaluate the biologic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study of beta-glucan.

Patients receive oral beta-glucan once daily on days -4 to 12 and monoclonal antibody 3F8 IV over 30-90 minutes on days 1-5 and 8-12. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity and with a human antimouse antibody (HAMA) titer < 1,000 U/mL.

Cohorts of 3-6 patients receive escalating doses of beta-glucan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients undergo urine, bone marrow, and blood sample collection periodically for biological studies. Samples are analyzed for antibody-dependent cellular cytotoxicity, complement-mediated cytotoxicity, and serum HAMA response via immunohistochemistry.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma by 1 of the following methods:

  * Histopathology
  * Bone marrow involvement AND elevated urinary catecholamines
* High-risk disease, defined by 1 of the following:

  * Stage 4 disease with MYCN amplification (any age) or without MYCN amplification (> 18 months of age)
  * MYCN-amplified stage 3 disease (unresectable and any age)
  * MYCN-amplified stage 4S disease
* Metastatic disease
* Tumor progression or persistent disease (at metastatic or primary site) after intensive conventional chemotherapy
* Must have evaluable (microscopic marrow metastasis, elevated tumor markers, positive MIBG or PET scans) or measurable (CT scan or MRI) disease documented after completion of prior systemic therapy

PATIENT CHARACTERISTICS:

* Platelet count > 25,000/mm^3
* ANC > 500/mm^3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergy to mouse proteins, beta-glucan, mushrooms, or yeast
* No active life-threatening infections
* No severe major organ toxicity

  * Concurrent toxicity must be ≤ grade 2 except for the following, which may be grade 3:

    * Myelosuppression
    * Hearing loss
    * Alopecia
    * Anorexia
    * Nausea
    * Hyperbilirubinemia from TPN
    * Anxiety
    * Hypomagnesemia
* No prior HAMA titer > 1,000 U/mL by ELISA

PRIOR CONCURRENT THERAPY:

* No concurrent supplemental beta-glucan in food (e.g., bran cereals or mushrooms) or as complementary medicine
* No other concurrent systemic anticancer medications (e.g., hormonal agents, chemotherapy, investigational agents, or immunotherapy)

  * Concurrent isotretinoin allowed after the second course of study treatment is completed or if the patient develops human antimouse antibody (HAMA)

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-09-09 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Toxicity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Brian H. Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Cardenas FI, Mauguen A, Cheung IY, Kramer K, Kushner BH, Ragupathi G, Cheung NV, Modak S. Phase I Trial of Oral Yeast-Derived beta-Glucan to Enhance Anti-GD2 Immunotherapy of Resistant High-Risk Neuroblastoma. Cancers (Basel). 2021 Dec 14;13(24):6265. doi: 10.3390/cancers13246265. PMID 34944886
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm